CLINICAL TRIAL: NCT03907657
Title: Double-Center Cross-Sectional Study of Contrast-Enhanced Ultrasound With Lumason/Definity as a Screening Tool for Kidney Cancer in Patients With Von-Hippel Lindau
Brief Title: Contrast-enhanced Ultrasound as a Screening Tool for Kidney Cancer in Patients With Von-Hippel Lindau
Acronym: CEUS-VHL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: Lantheus Medical Imaging (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: LCCC1824
Record Dates: First submitted 2019-04-05; First posted 2019-04-09 (Actual); Results first posted 2024-05-21 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Von-Hippel Lindau; Kidney Disease, Chronic
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — perflutren

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Perflutren Lipid Microsphere or Lumason (Experimental): Patients with Von-Hippel Lindau disease will be imaged using contrast-enhanced ultrasound with either perflutren or Lumason.
  Interventions: Drug: Perflutren lipid microsphere; Drug: Sulfur hexafluoride lipid microspheres

INTERVENTIONS:
Drug: Perflutren lipid microsphere — Baseline B-mode US will be performed to confirm the lesions being imaged (unless it is a subject with no lesions, then a basic B-mode US will be performed. Perflutren is a diagnostic drug that is intended to be used for contrast enhancement. The vial contains a clear, colorless, sterile, non-pyrogenic, hypertonic solution which is activated by mechanical agitation with Vialmix®.It will be dispensed in inactivated form to a study team member. The contrast agent will be activated just prior to administration (ideally to be used within 5 minutes of activation). Contrast agent Definity (or Lumason) will be activated according to package insert instructions, including use of VialMix®, the device used to activate Definity. Administration will occur IV in coordination with sonography staff trained specifically in contrast ultrasound imaging.The total imaging time is anticipated to be less than 30 minutes.
  Other Names: • Definity®; • Microbubble contrast agent
Drug: Sulfur hexafluoride lipid microspheres — Baseline B-mode US will be performed to confirm the lesions being imaged (unless it is a subject with no lesions, then a basic B-mode US will be performed. Lumason will be used as a secondary contrast agent only if Definity(perflutren) is unavailable.This drug will be administered using the dosing range and administration type within the Lumason prescribing information. The contrast agent will be activated just prior to administration (ideally to be used within 5 minutes of activation). Contrast agent Definity (or Lumason) will be activated according to package insert instructions, including use of VialMix®, the device used to activate Definity. Administration will occur IV in coordination with sonography staff trained specifically in contrast ultrasound imaging.The total imaging time is anticipated to be less than 30 minutes.
  Other Names: Lumason

SUMMARY:
The purpose of this study is to determine if contrast-enhanced ultrasound can detect abnormal features of kidney lesions in patients with Von-Hippel Lindau with the same accuracy as conventional ultrasound and contrast-enhanced magnetic resonance imaging (MRI)

DETAILED DESCRIPTION:
This is a pilot cross-sectional study that compares contrast enhanced ultrasound to conventional ultrasound and contrasted MRI. Any patient undergoing annual imaging screening is eligible, but the investigators will target inclusion of at least 10 subjects who have at least 1 kidney lesion. Therefore, up to 5 subjects may have no current kidney lesions. Subject participation will be only for the day of CEUS study. There will be no follow-up period for this study. However, if results are encouraging, a longitudinal observational study may follow, and these same subjects would be eligible for enrollment. Eligible subjects will undergo a contrast enhanced ultrasound.

Following completion of imaging, all CEUS, MRI (within 4 months) and B-mode (at time of CEUS) US studies will be de-identified. Blinded radiologists will interpret images and provide an overall assessment of risk of malignancy to each kidney using the Bosniak criteria for each kidney lesion present. The Bosniak criteria places cystic lesions into one of 5 categories (I, II, IIF, III and IV) based on lesion characteristics. CEUS based diagnosis will be compared to the diagnoses on routine B-mode US and contrast-enhanced MRI.

ELIGIBILITY:
Inclusion Criteria:

To be eligible for the present study, patients must meet the following criteria:

1. Able to provide written informed consent
2. Willing to comply with protocol requirements
3. At least 16 years of age
4. Carry a diagnosis of VHL and able to undergo routine clinical screening tests for RCC

Exclusion Criteria:

1. Critically ill or medically unstable or in an intensive care setting and whose critical course during the observation period would be unpredictable
2. Known hypersensitivity to sulfur hexafluoride or to any component of perflutren lipid (Definity®) or sulfur hexafluoride (Lumason®)
3. Right to left shunt, severe pulmonary hypertension (Pulmonary artery pressure >90mmHg), or adult respiratory distress syndrome
4. Active cardiac disease including any of the following:

   A. Severe congestive heart failure (class IV in accordance with the classification of the New York Heart Association) B.Unstable angina. C.Symptomatic arrhythmia (i.e. tachycardia, bradycardia, supraventricular tachycardia, ventricular fibrillation, ventricular tachycardia, atrial flutter or fibrillation).

   D.Myocardial infarction within 14 days prior to the date of proposed microbubble administration.
5. Has any other medical condition or other circumstances that would significantly decrease the chances of obtaining reliable data or of achieving the study objectives such as:

   * Mental illness
   * Drug abuse
6. Female patient who is pregnant or lactating
7. Obesity that limits obtainment of acceptable images

Ages: 16 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2019-09-23 (Actual); Primary Completion 2023-03-13 (Actual); Study Completion 2023-03-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emily Chang, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina of Chapel hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Larcher A, Rowe I, Belladelli F, Fallara G, Raggi D, Necchi A, Montorsi F, Capitanio U, Salonia A; OSR VHL Program. Von Hippel-Lindau disease-associated renal cell carcinoma: a call to action. Curr Opin Urol. 2022 Jan 1;32(1):31-39. doi: 10.1097/MOU.0000000000000950. PMID 34783716

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Subjects were enrolled in one center in North Carolina, between 9/23/2019 - 02/13/2023. All considered subjects were eligible, consented, and completed the study. In total 29 kidneys were studied.
Groups:
- All Subjects: All Patients with genetic diseases at risk of kidney lesions.
Period: Overall Study Subjects
Arm/Group | All Subjects
Started | 15
Completed | 15
Not Completed | 0
Period: CEUS
Arm/Group | All Subjects
Started | 15
Completed | 15
Not Completed | 0
Period: B Mode
Arm/Group | All Subjects
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Patients with a genetic disease at risk of kidney lesions will be imaged using contrast-enhanced ultrasound with Perflutren and their clinical MRI images performed within 4 months.
Groups:
- Patients With a Genetic Disease at Risk of Kidney Lesions: Patients with a genetic disease at risk of kidney lesions will be imaged using contrast-enhanced ultrasound with Perflutren.
Arm/Group | Patients With a Genetic Disease at Risk of Kidney Lesions
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 15
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 15
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 12
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Comparison in Radiologist's Lesion Evaluation: CEUS Versus B-mode Ultrasound
Description: Each reader will evaluate kidney imaging using Contrast-Enhanced Ultrasound (CEUS) versus Brightness Mode Ultrasound (B-mode) in patients at risk for kidney lesions. A dichotomized Bosniak score was used for comparison. Dichotomized Bosniak score: 0= nonmalignant and 1=malignant or possibly malignant. Scores were averaged across all readers. Kidneys were assessed by CEUS and B-mode by three different readers.
Time Frame: Baseline
Population: Patients with a genetic disease at risk of a kidney lesion were imaged using contrast-enhanced ultrasound with Perflutren and B-mode ultrasound. Twenty- nine kidneys belonging to fifteen patients were assessed.
Measure: Mean (Full Range); unit: Dichotomized score
Units Other Than Participants: Overall Number of Kidneys
Groups:
- CEUS: Contrast-enhanced ultrasound (CEUS) technique was used to evaluate 29 kidneys belonging to 15 subjects.
- B-Mode: Brightness Mode Ultrasound (B-mode) technique was used to evaluate 29 kidneys belonging to 15 subjects.
Arm/Group | CEUS | B-Mode
Number analyzed (Participants) | 15 | 15
Number analyzed (Overall Number of Kidneys) | 29 | 29
Dichotomized score | 0.13 [0 to 1] | 0.20 [0 to 1]

2. Secondary Outcome: Comparison in Radiologist's Lesion Evaluation: CEUS Versus Clinically Performed MRI
Description: Each reader will evaluate kidney imaging using Contrast-Enhanced Ultrasound (CEUS). Potentially malignant lesions were extracted from clinically performed magnetic resonance imaging (MRI) completed within 4 months of CEUS. Dichotomized Bosniak scores from CEUS were compared with MRI-derived malignancy scores.
  Dichotomized Bosniak scores: 0= nonmalignant and 1=malignant or possibly malignant. Scores were averaged across all readers.
Time Frame: Baseline
Population: Patients with a genetic disease at risk of kidney lesions will be imaged using contrast-enhanced ultrasound with Perflutren.Twenty- nine kidneys belonging to fifteen patients were assessed.
Measure: Mean (Full Range); unit: Dichotomized score
Units Other Than Participants: Overall Number of Kidneys
Groups:
- Magnetic Resonance Imaging: Magnetic Resonance Imaging was used to evaluate 29 kidneys belonging to 15 subjects.
Arm/Group | CEUS | Magnetic Resonance Imaging
Number analyzed (Participants) | 15 | 15
Number analyzed (Overall Number of Kidneys) | 29 | 29
Dichotomized score | 0.13 [0 to 1] | 0.10 [0 to 1]

ADVERSE EVENTS:
Time Frame: Up to 1 day
Description: Adverse events were collected from day one of the study contrast agent administration.
Arm/Group | Patients With a Genetic Disease at Risk of Kidney Lesions
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-01-18): https://cdn.clinicaltrials.gov/large-docs/57/NCT03907657/Prot_SAP_000.pdf